CLINICAL TRIAL: NCT01944917
Title: Pilot Study to Investigate Autonomic Function in Patients With Chronic Musculoskeletal Pain.
Brief Title: Effects of Pulsed Electromagnetic Field on Autonomic Function in Patients With Chronic Musculoskeletal Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aerotel Ltd (Industry)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: DGS2013
Record Dates: First submitted 2013-08-25; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Musculo-skeletal Pain
Keywords: Electromagnetic field; VAS score; Heart Rate Variability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic musculoskeletal pain: Chronic musculoskeletal pain - treated with electromagnetic field Chronic musculoskeletal pain - placebo

SUMMARY:
Previously it has been demonstrated that exposing the heart to electromagnetic field during exercise stress test improves the recovery following the stress test. This is explained by the effect of the electromagnetic field on the sympathetic activity of the heart. In the present study we would like to further investigate the effects of electromagnetic field on autonomic nervous system function in patients with chronic musculoskeletal pain that usually have high sympathetic activity. Each patient will be exposed to 20 minutes of electromagnetic field during which the autonomic nervous system function will be measured. In addition, patient tolerability to the exposed magnetic field will be investigated. We assume that short exposure to electromagnetic field would result in decreased sympathetic activity and therefore, on the long run, could be suggested as a therapeutic tool for such patients.

DETAILED DESCRIPTION:
Adult patients suffering from chronic muscoloskeletal pain will be recruited to this study during their weekly visits to the Department for Complementary Medicine at Sheba Medical Center. Patient will be exposed to 20 minutes of weak intensity and low frequency electromagnetic field while seated, during which heart rate variability measures will be recorded. In addition, patient tolerability to the exposed electromagnetic field will be investigated, including VAS score (pain score). This is a double blind placebo-control study by which neither the patients nor the physicians know which treatment is given to the patients. The study code will be open only at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Chronic musculoskeletal pain

Exclusion Criteria:

* Implantable defibrillator
* Implantable pacemaker
* Active cancer
* Pregnancy

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from musculoskeletal pain visiting weekly the Department for Complementary Medicine at Sheba Medical Center will be recruited to this study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Reduced heart rate variability measures associated with sympathetic activity | By the end of the experiment: following 20 minutes of PEMF exposure.
  Heart rate variability will be measured at baseline, prior to exposure to PEMF, and continuously for 20 minutes during exposure to PEMF, and 5 minute thereafter, after removal of the PEMF. Changes in heart rate variability (increase in high frequency and decrease in low frequency spectra) between exposure to PEMF and baseline will be evaluated. We hypothesize that heart rate variability measures reflecting sympathetic activity (low frequency spectra) will be reduced during exposure to PEMF with consequence increase in parasympathetic autonomic activity (high frequency spectra).

SECONDARY OUTCOMES:
Reduced VAS score | Immediately at the end of the experiment: following 20 minutes of PEMF exposure.
  Since VAS is visual analogue scale pain score that reflects sympathetic activity we expect to monitor a reduced score following exposure to PEMF, which should be in correlation with increased parasympathetic activity (as measured by heart rate variability measures).

OTHER OUTCOMES:
No change in patients tolerability to the electromagnetic field | Immediately at the end of the exposure: following 20 minutes of PEMF exposure.
  As a secondary outcome we would like to assess patients tolerability to 20 minutes exposure to PEMF. We do not expect any change in tolerability score due to the exposure to PEMF.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Complementary Medicine, Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Result] Grote V, Lackner H, Kelz C, Trapp M, Aichinger F, Puff H, Moser M. Short-term effects of pulsed electromagnetic fields after physical exercise are dependent on autonomic tone before exposure. Eur J Appl Physiol. 2007 Nov;101(4):495-502. doi: 10.1007/s00421-007-0520-x. Epub 2007 Aug 3. PMID 17674028